CLINICAL TRIAL: NCT01498016
Title: Pharmacokinetic Study of Intravenous Busulfan as Conditioning Regimen for Allogeneic Stem Cell Transplantation in Adult Patients With Acute Leukemia
Brief Title: Pharmacokinetic Study of Busulfan in Allogeneic Stem Cell Transplantation in Adult Patients With Acute Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood &^ Marrow Transplantation Center, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJH-Busulfan
Record Dates: First submitted 2011-12-19; First posted 2011-12-23 (Estimated); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Acute Leukemia
Keywords: acute leukemia; allogeneic stem cell transplantation; busulfan
MeSH Terms: interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iv-Busulfan (Experimental): iv busulfan 1.6mg/kg given q12h
  Interventions: Drug: Busulfan

INTERVENTIONS:
Drug: Busulfan — Iv busulfan 1.6mg/kg q12h D1- D4
  Other Names: study group

SUMMARY:
Intravenous Busulfan (iv-Bu) is commonly used as part of preparation regimen for allogeneic hematopoietic stem cell transplantation for patients with acute leukemia. Though the pharmacokinetics data are available for population from America, Europe and Japan or Korea in Asia, there are no data in Chinese population. It is shown that high Bu concentration are associated with the toxicity such as veno-occlusion disease and lower concentration is correlated with reduced anti-leukemia effect, thus the monitoring of Bu and/or the strategy to achieve an optimal target Bu concentration are accepted to avoid toxicity while maintain the anti-leukemia effect which may overall improve the outcome of allo-SCT. Thus we conduct the pharmacokinetic study in Chinese population.

DETAILED DESCRIPTION:
All patients received intravenous Busulfan based conditioning regimen for allogeneic stem cell transplantation.

Intravenous Busulfan (iv-Bu) was given 1.6mg/kg twice daily for 4 days as in the conditioning regimen.

Blood samples were obtained after first and 7th dose of iv Bulsulfan.

ELIGIBILITY:
Inclusion Criteria:

* patient with acute myeloid or lymphoblastic leukemia in 1st or second remission
* age 18-55 years
* with inform consent
* no contraindication for allogeneic transplantation: active infection, allergy to FLu/Bu/CTX, liver and renal function damage
* HLA matched related (6/6) or unrelated donors (at least 8/10)

Exclusion Criteria:

* age less than 18 years or over 56 years
* HLA mismatched related donor
* liver function/renal function damage (over 2 X upper normal range)
* with mental disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-11; Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | predose, 0,1,2,3,4,6,8,12,24,48,72, 96 hours post-dose
  busulifan blood concentration

CONTACTS AND LOCATIONS:
Overall Officials: Jiong HU, M.D., Principal Investigator — Rui Jin Hospital, Shanghai JiaoTong University School of Medicine
Locations (1):
- Blood & Marrow Transplantation Center, RuiJin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No